CLINICAL TRIAL: NCT00000995
Title: Phase I Studies of the Combination of AZT and DHPG (Ganciclovir) in Patients With AIDS and Cytomegalovirus Infection
Brief Title: A Study of AZT Plus Ganciclovir in Patients With AIDS and Cytomegalovirus (CMV) Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 004; 10980 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Cytomegalovirus Infections; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Ganciclovir; Drug Evaluation; Drug Therapy, Combination; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — Cytomegalovirus Infections; HIV Infections; AIDS-Related Opportunistic Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Acquired Immunodeficiency Syndrome | interventions — Zidovudine; Ganciclovir

INTERVENTIONS:
Drug: Zidovudine
Drug: Ganciclovir

SUMMARY:
To evaluate the clinical and laboratory toxicity of ganciclovir (GCV) and zidovudine (AZT) when given in combination.

Because recent information has shown AZT to be useful in treating AIDS, it is assumed that most patients with AIDS, and probably with AIDS related complex (ARC), will be receiving AZT. Because AZT is reported not to be active against cytomegalovirus (CMV), it is important to see if it is useful to give GCV along with AZT.

DETAILED DESCRIPTION:
Because recent information has shown AZT to be useful in treating AIDS, it is assumed that most patients with AIDS, and probably with AIDS related complex (ARC), will be receiving AZT. Because AZT is reported not to be active against cytomegalovirus (CMV), it is important to see if it is useful to give GCV along with AZT.

Patients are placed into one of four groups at entry into study according to their previous treatment:

I: Prior treatment with AZT up to the time of developing CMV infection and not requiring dose reduction of AZT for toxicity.

II: Prior treatment with AZT up to the time of developing CMV infection and requiring dose reduction of AZT for toxicity.

III: Prior therapy with GCV for CMV infection. These patients should already be in the maintenance phase, having completed a minimum of 2 weeks of induction therapy.

IV: No prior therapy with either AZT or GCV.

Treatment lasts 24 weeks and consists of two treatment plans:

A: Patients not previously treated with GCV are started on GCV for an additional 22 weeks. GCV is given as a 1-hour infusion. All patients are started on AZT at the lowest dose. B: For patients with chronic CMV disease who are receiving GCV maintenance, GCV is administered as a 1-hour infusion 5 days/week.

AZT is added and treatment with GCV is standardized prior to beginning of the study.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Symptomatic therapy such as analgesics, antihistamines, antiemetics, and antidiarrheal agents, or other supportive therapy may be administered as deemed necessary by the responsible investigator. For fever, the following regimens should be used:
* If fever above 39.0 degrees C, antipyretic therapy will be administered employing aspirin, 650 mg orally every 4 hours x 3 doses, or until fever falls below 39.0 degrees C.
* If fever of higher than 39.0 degrees C occurs for 2 consecutive days, the patient may be premedicated with aspirin.

Exclusion Criteria

* Active alcohol or drug abuse.

Co-existing Condition:

Excluded:

* Patients with other life-threatening and uncontrolled opportunistic infections on enrollment.

Patients with the following prior conditions are excluded if they:

* Have other life-threatening and uncontrolled opportunistic infections on enrollment.

Prior Medication:

Excluded within 1 week of study entry:

* Systemic therapy with antimetabolite.
* Cytotoxic drug.
* Interferon.
* Immunologic modulators.
* Corticosteroids.
* Nucleoside analogs other than zidovudine (AZT).
* Excluded within 2 weeks of study entry:
* Therapy for any other opportunistic infections.
* Excluded within 2 months of study entry:
* Ribavirin.

Prior Treatment:

Excluded within 2 weeks of study entry (for treatment group I):

* Blood transfusion.
* Excluded within 1 month of study entry (for treatment groups II and III):
* Blood transfusion.

All patients must be:

* Able to provide informed consent.
* Likely to be available for follow-up for at least 4 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Study Completion 1990-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reichman RC, Study Chair; Richman D, Study Chair; Hochster H, Study Chair
Locations (3):
- United States (3):
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York

REFERENCES:
- [Background] Hochster H, Dieterich D, Bozzette S, Reichman RC, Connor JD, Liebes L, Sonke RL, Spector SA, Valentine F, Pettinelli C, et al. Toxicity of combined ganciclovir and zidovudine for cytomegalovirus disease associated with AIDS. An AIDS Clinical Trials Group Study. Ann Intern Med. 1990 Jul 15;113(2):111-7. doi: 10.7326/0003-4819-113-2-111. PMID 2163228